CLINICAL TRIAL: NCT04610411
Title: Evaluation of the Accuracy of Surgical Navigation in Spine Instrumentation Using Augmented Reality
Acronym: HoloNavi
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Balgrist University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: HoloNavigation
Record Dates: First submitted 2020-06-08; First posted 2020-10-30 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2023-02

CONDITIONS: Surgery
MeSH Terms: interventions — Surgery, Computer-Assisted

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- surgical navigation (Experimental): standard surgical method except for navigated instrumentation of pedicle screws and rod implants
  Interventions: Device: surgical navigation
- standard surgical method (Active Comparator): standard surgical method established at the institution
  Interventions: Other: standard surgical method

INTERVENTIONS:
Device: surgical navigation — surgical navigation for pedicle screw placement and rod beinding using AR-glasses and a specially developed software
  Arms: surgical navigation
Other: standard surgical method — standard surgical method established at the institution
  Arms: standard surgical method

SUMMARY:
This study will investigate the accuracy of implant navigation for spinal instrumentation. The tested technique is based on commercially available AR-glasses and a specially developed software component

DETAILED DESCRIPTION:
The experimental intervention consists of using the AR-glasses and a specially developed software as a navigation aid in surgery. The surgical technique for the intervention group corresponds to the established standard method. It is identical to the control intervention except for the step where pedicle screws or rod implants are instrumented.

The surgeon wears the hardware component during the entire surgery. He proceeds conventionally up to the point where navigation of pedicle screws and rod implants with is required.

ELIGIBILITY:
Inclusion Criteria:

* Indication for surgical instrumentation of the spine (Os Sacrum, L1-L5, Th1-Th12) without or with correction of a malposition.
* Anatomical adaptation of the rod implant necessary.
* The trial participant is able to give his/her consent.
* Signed written declaration of consent after oral and written explanation.
* Male and female patients aged 18 years and older.
* Indication for a preoperative CT scan of the lumbar spine
* Existence of a preoperative planning, which was created on the basis of 3D CT imaging

Exclusion Criteria:

* Pregnant or breastfeeding women
* Emergency situations
* Other known clinically significant concomitant diseases (e.g. infections, tumors, co-existing arthrosis).
* Known or suspected incompliance with the protocol, such as drug or alcohol abuse.
* Inability of the patient to follow the study procedures, e.g., due to language problems, mental illness, dementia, etc.
* There is no conventional surgical treatment that can be used if the MP cannot be used intraoperatively.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2024-04-11 (Actual); Study Completion 2024-04-12 (Actual)

PRIMARY OUTCOMES:
Accuracy | within 7 days of surgery
  3-dimensional deviation (3D angle) of preoperative planning in postoperative imaging
Accuracy | within 7 days of surgery
  3-dimensional deviation (3D translation vector) of preoperative planning in postoperative imaging

SECONDARY OUTCOMES:
Number of rod bending attempts | during surgery
  bending attempts are counted during surgery
Number of length corrections of rod implant | during surgery
  required length corrections are counted during surgery
time needed for pedicle screw implantation | during surgery
  time is measured during surgery
surgery duration | during surgery
  total Duration of surgery
Radiation dose during surgery | during surgery
  total radiation dose applied during surgery
Usability | within 7 days of surgery
  measuring of surgeon satisfaction using visual analogue scale from a minimum of 0 to a maximum of 10
Clinical Outcome Pain | up to 1 year of surgery
  Standardized clinical pain score (visual analogue scale for pain with 0=no pain and 10=unbearable pain) is routinely evaluated before surgery and in the follow up
Clinical Outcome Disability | up to 1 year of surgery
  Standardized clinical disability score (Oswestry Low Back Pain Questionnaire with 0%=minimal disability and 100%=maximal disability ) is routinely evaluated before surgery and in the follow up

CONTACTS AND LOCATIONS:
Overall Officials: Mazda Farshad, Prof., Principal Investigator — Balgrist University Hospital
Locations (1):
- Balgrist University Hospital, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No